CLINICAL TRIAL: NCT05949619
Title: A Phase Ib/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BL-M02D1 for Injection in Patients With Multiple Solid Tumors, Including Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of BL-M02D1 in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer or Other Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M02D1-103
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-M02D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M02D1

INTERVENTIONS:
Drug: BL-M02D1 — Administration by intravenous infusion

SUMMARY:
Phase Ib: To explore the safety and preliminary efficacy of BL-M02D1 to further define RP2D in a variety of solid tumors such as locally advanced or metastatic non-small cell lung cancer. Phase II: To explore the efficacy of BL-M02D1 using single-agent RP2D obtained from phase I clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. No gender limit;
3. Age: ≥18 years old;
4. expected survival time ≥3 months;
5. Histologically and/or cytologically confirmed locally advanced or metastatic non-small cell lung cancer and other solid tumors that have failed standard treatment;
6. Consent to provide archival tumor tissue specimens (10 unstained sections (anti-slip) surgical specimens (thickness 4-5μm)) or fresh tissue samples from primary or metastatic lesions within 3 years. If participants cannot provide tumor tissue samples, they can be enrolled if they meet other inclusion and exclusion criteria, after the evaluation of the investigator;
7. Must have at least one measurable lesion according to RECIST v1.1 definition;
8. ECOG 0 or 1;
9. Toxicity from previous antineochemical therapy has returned to grade 1 or less as defined by NCI-CTCAE v5.0 (asymptomatic laboratory abnormalities such as elevated ALP, hyperuricemia, elevated serum amylase/lipase, and elevated blood glucose were considered by the investigator, and toxicity with no safety risk was judged by the investigator; Excluding alopecia, grade 2 peripheral neurotoxicity, hypothyroidism stabilized by hormone replacement therapy, or decreased hemoglobin (≥90g/L).
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. The level of organ function must meet the following requirements and meet the following standards:

    1. Bone marrow function: absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥90 g/L;
    2. Liver function: total bilirubin (TBIL≤1.5 ULN), AST and ALT ≤2.5 ULN in patients without liver metastasis, AST and ALT ≤5.0 ULN in patients with liver metastasis;
    3. Renal function: creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to Cockcroft and Gault formula).
12. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5ULN;
13. Urine protein ≤2+ or ≤1000mg/24h;
14. Female subjects of childbearing potential or male subjects with a fertile partner must use highly effective contraception from 7 days before the first dose until 6 months after the dose. Female subjects of childbearing potential had to have a negative serum pregnancy test within 7 days before the first dose.

Exclusion Criteria:

1. Antineoplastic therapy, including chemotherapy, biologic therapy, immunotherapy, definitive radiotherapy, major surgery (investigator-defined), or targeted therapy (including small-molecule tyrosine kinase inhibitors), has been administered within 4 weeks or 5 half-lives (whichever is shorter) before the first dose; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Oral fluorouracil drugs such as S-1, capecitabine, or palliative radiotherapy within 2 weeks before the first dose; The TCM with anti-tumor indications was within 2 weeks before the first administration.
2. Prior treatment with Trop2-targeted ADC drugs or with camptothecin derivatives (topoisomerase I inhibitors) as toxins;
3. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

   1. severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, third degree atrioventricular block, complete left bundle branch block, frequent and uncontrollable arrhythmias, such as atrial fibrillation, atrial flutter, ventricular fibrillation, and ventricular flutter (except transient);
   2. prolonged QT interval at rest (QTc > 450 msec in men or QTc > 470 msec in women);
   3. acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before the first dose;
   4. patients with New York Heart Association (NYHA) functional class ≥II heart failure;
4. Patients at risk for active autoimmune disease, or with a history of autoimmune disease, Including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener syndrome, autoimmune hepatitis, systemic sclerosis, Hashimoto's thyroiditis, autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome), etc. Exceptions were type I diabetes, hypothyroidism that was stable with hormone-replacement therapy (including that due to autoimmune thyroid disease), psoriasis or vitiligo that did not require systemic therapy, and hypothyroidism that was stable with hormone-replacement therapy.
5. Patients with other malignant tumors within 5 years before the first administration, except those who have been cured skin squamous cell carcinoma, basal cell carcinoma, superficial bladder cancer, prostate/cervix/breast cancer in situ and so on are considered to be eligible for enrollment;
6. Unstable deep vein thrombosis, arterial thrombosis, and pulmonary embolism requiring medical intervention within 6 months before screening; Infusion-related thrombosis was excluded.
7. Patients with massive or symptomatic effusions, or poorly controlled effusions (poorly controlled was defined as requiring 2 or more paracentesis within a month).
8. Hypertension poorly controlled by two antihypertensive drugs (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
9. Current interstitial lung disease, drug-induced interstitial pneumonia, radiation pneumonitis requiring steroid therapy, or a history of these diseases;
10. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (meningeal metastases). Patients who had received treatment for brain metastases (radiotherapy or surgery; Patients with stable brain metastases who had stopped radiotherapy or surgery 28 days before the first dose were eligible. Patients with cancerous meningitis (meningeal metastasis) were excluded even if they were treated and judged to be stable. Stable disease was defined as being asymptomatic, in stable condition, and not requiring steroid therapy for more than 4 weeks before starting study treatment.
11. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or any of the excipients of BL-M02D1;
12. Previous history of allogeneic stem cell, bone marrow, or organ transplantation;
13. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBsAg positive or HBcAb positive and HBV-DNA copy number > central detection lower limit) or hepatitis C virus infection (HCV antibody positive and HCV-RNA > central detection lower limit);
14. Severe systemic infection occurred within 4 weeks before screening, including but not limited to severe pneumonia caused by fungi, bacteria, viruses, bacteremia, or serious infectious complications;
15. A history of autologous or allogeneic stem cell transplantation;
16. Pregnant or lactating women;
17. Other conditions for participation in the trial were not considered appropriate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Recommended Phase II Dose (RP2D) | Up to 21 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M02D1.
Phase II: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M02D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M02D1.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase II: Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-M02D1 to the first date of either disease progression or death, whichever occurs first.
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of BL-M02D1 will be investigated.
Tmax | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of BL-M02D1 will be investigated.
Ctrough | Up to 21 days after the first dose
  Ctough is defined as the lowest serum concentration of BL-M02D1 prior to the next dose will be administered.
Phase Ib: T1/2 | Up to 21 days after the first dose
  Half-life (T1/2) of BL-M02D1 will be investigated.
Phase Ib: AUC0-T | Up to 21 days after the first dose
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
Phase Ib: CL | Up to 21 days after the first dose
  CL in the serum of BL-M02D1 per unit of time will be investigated.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-M02D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, PHD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China